CLINICAL TRIAL: NCT05812690
Title: An International Study of Molar Incisor Hypomineralisation and Its Association With Dental Anomalies
Brief Title: Molar Incisor Hypomineralisation and Dental Anomalies
Status: Completed | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH21833
Record Dates: First submitted 2023-03-31; First posted 2023-04-14 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Molar Incisor Hypomineralisation
Keywords: Molar Incisor Hypomineralisation; Dental Anomalies; Children; Hypodontia
MeSH Terms: conditions — Molar Hypomineralization; Tooth Abnormalities; Anodontia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with molar incisor hypomineralisation: Children referred to the host centres with a clear diagnosis of MIH, as given by a specialist paediatric dentist
  Interventions: Other: This is a non intervention - observation only study
- Children without molar incisor hypomineralisation: Children referred to the host centres with no evidence of MIH
  Interventions: Other: This is a non intervention - observation only study

INTERVENTIONS:
Other: This is a non intervention - observation only study — This is non intervention study

SUMMARY:
Background/study aim:

Molar incisor hypomineralisation (MIH) is a common disorder of tooth development. Affected teeth have weak enamel and adult molars often require extensive treatment or even extraction. A preliminary study, carried out in Sheffield Dental Hospital, discovered that 12% of MIH children also had congenitally missing adult teeth, presenting further challenges to treatment-planning. This novel finding stimulated discussion between international MIH experts; whilst some clinicians had observed this association, others had not. Therefore the primary aim of this international study is to determine the association between MIH and missing teeth in different populations. This has important clinical and biological relevance in understanding the presentation and management of MIH.

Participants/research sites:

This study will include 584 children with MIH and a comparison group of 584 children without MIH. Young dental patients, aged 7-16 years, who attend for a check-up or treatment at one of the 15 participating countries will be invited to take part. The UK sites are Sheffield, Newcastle and University College London Dental Hospitals and all children will be seen by specialists/consultants in paediatric dentistry to confirm their diagnosis of MIH. The main inclusion criteria is that children have a dental xray as part of their routine care.

Data collection:

Following a routine dental check-up we will grade the severity of the participants' MIH (if present) and record any other dental anomalies (e.g. abnormal tooth number, position or shape). We will also check the dental xray for other anomalies that cannot be seen from the clinical exam. We will analyse the prevalence of MIH and association with other dental anomalies to see if there are difference according to sex or ethnicity and compare our findings with the non-MIH group. We anticipate the study will take 18 months.

DETAILED DESCRIPTION:
The primary objective is to compare the overall prevalence of congenitally missing teeth/hypodontia (excluding wisdom teeth) in children (7-16 years old) with and without MIH.

Secondary research questions/objectives

The secondary research objectives are to:

1. Compare the prevalence of developmentally missing teeth (hypodontia) in MIH children based on region, ethnicity and gender
2. Determine the clinical pattern (including symmetry), severity and treatment need of MIH in children (aged 7-16years) referred to specialist paediatric dentistry services across the world, according to gender and ethnic group/region
3. Compare the prevalence of other co-existing developmental dental anomalies between the two groups
4. Compare the prevalence of developing third permanent molars between the two groups

What is the scientific justification for the research?

Molar incisor hypomineralisation (MIH) is one of the most common disorders of tooth development seen in paediatric dentistry practice around the world. A recent meta-analysis of 99 studies, in 43 different countries, estimated the global prevalence of MIH to be 13.1% with significant variations seen between super-regions, regions and countries.

A wide variety of other dental anomalies are also seen in childhood, broadly encompassing deviations in tooth number, morphology, structure, position and eruption. Prevalence data for all these different developmental disorders vary widely, depending on the anomaly in question, diagnostic approach and the target population . It is also important to note that the presence of one anomaly should always alert clinicians to the possibility of others, as numerous studies have demonstrated significant inter-relationships between certain anomaly types. Recently, a UK study explored, for the first time, the prevalence of dental anomalies in children diagnosed with MIH. Clinical and radiographic examination of 101 children aged 6-15 years found that, in total, 29% of patients had another dental anomaly in addition to MIH (Walshaw et al., 2020).

There are established guidelines for the management of children with MIH. In some situations, the extraction of one or more first permanent molars is the preferred option, providing all other permanent teeth (and preferably third permanent molars/wisdom teeth) are present. Thus, the congenital absence of a second premolar in the same quadrant would have considerable impact on this decision and potentially compromises long-term outcomes. A controlled study, exploring any association between the presence of MIH and hypodontia, in addition to other dental anomalies, is clearly warranted to better inform patient management. The need for earlier radiographic examination and definitive treatment for hypomineralised first permanent molars would be paramount if such an association is confirmed by the proposed multi-centre international study.

Design and methodology.

This will be a cross-sectional study involving children with MIH and a comparison group of non MIH-affected children.

Burden to research participants Research participants (MIH and comparison group) will not be required to attend any additional visits other than their scheduled check-up or treatment visit. However, their dental check up will take slightly longer than normal (around an extra 5 minutes) as we will be recording in more detail than usual the condition of their enamel (using a validated scoring system of MIH). They will have a dental xray taken as part of their 'routine care' so will not be exposed to unnecessary ionising radiation. They will also be invited to have clinical photographs of their teeth, which may not have been part of their 'routine care'. They will also be verbally asked two (validated) questions about how they rate their own oral health, which is not part of routine care.

Study population

Participants will be recruited from patients attending for treatment, a recall or new patient assessment, in the host centres. Written informed consent will be obtained for study participation from parents/guardians and children. The 'experimental ' group will be children aged 7-16 years referred to specialist paediatric dentistry services for the management of MIH in the following countries:

1. Nigeria
2. Australia-2 centres (both Melbourne)
3. Chile
4. Egypt
5. India
6. Jordan
7. Netherlands- 2 centres
8. New Zealand
9. Qatar
10. Singapore
11. South Sudan
12. United Kingdom- 3 centres (London, Newcastle, Sheffield)
13. United States of America
14. United Arab Emirates
15. Saudi Arabia

A sample size of 1168 children (584 per group) was calculated. In order to achieve this sample size, each centre will aim to recruit 84 participants (42 patients per MIH group and 42 patients per control group).

Examiner training and calibration

Examiner training and calibration will be conducted on-line, using Microsoft Teams, using a set of ten clinical images and radiographs to ensure that there is acceptable intra-and inter-examiner agreement for key parameters under investigation as follows:

* Use of a validated MIH index to record severity status for first permanent molars;
* Clinical and radiographic diagnosis of all dental anomalies (abnormal tooth size, position and shape)
* Presence/absence of developing third permanent molars (wisdom teeth)
* Degree of taurodontism (this is an abnormal root canal shape) in lower first permanent molars using established criteria/index All clinicians involved in recording these parameters will have to reach acceptable levels of repeatability.

Examination and data collection An electronic data collection 'form' will be developed and piloted prior to commencement of the main study. The following non-identifiable patient and clinical variables will be recorded prior to transfer to a shared electronic dataset using secure processes.

Demographics

* Age
* Sex
* Ethnicity
* Primary dental diagnosis for both MIH and control participants.
* Children's global assessment of their own oral health status Radiographic characteristics All participants must have a full panoral (dental) radiograph of good diagnostic quality, taken for 'routine care'. A record will be made of any abnormalities of tooth shape, number and position from the radiographic presentation.

Assessment of taurodontism (abnormal root canal shape) For patients with mature apical development of their first permanent mandibular molars (10 years and over) an objective assessment of taurodontism will be carried out using digital measurements from panoral (dental) radiographs. This will be done according to established protocols; in brief, a diagnosis of taurodontism will be made if the crown/root ratio of the tooth is >1.1 (indicating that the crown pulp shape is abnormally elongated compared to the root length).

Data entry and statistical analysis.

Each unit will be responsible for anonymised electronic data entry for their participants and will send the complete data set securely to the principal investigators for data analysis.

Simple descriptive analysis will be used to present the demographic, clinical and radiographic findings for the MIH and control groups. In addition, statistical tests will be applied to determine:

* Any significant difference in the prevalence of dental anomalies (notably congenitally missing teeth) between children with and without a diagnosis of MIH and according to gender and ethnicity
* Any significant difference in the prevalence/degree of taurodontism (abnormal root canal shape) between children with and without a diagnosis of MIH and according to gender and ethnicity
* Any significant associations between the severity of MIH and presence of developing wisdom teeth, taurodontism and dental anomalies, according to gender and ethnicity

ELIGIBILITY:
Eligibility criteria Participants are children aged 7-16 years-old, with and without MIH, who meet the inclusion criteria, and attend for assessment or treatment in the participating clinics. To avoid bias, the comparison group will not be solely drawn from a pool of orthodontic patients or those primarily referred with a known diagnosis of dental anomalies

Generic inclusion criteria - all participants (both MIH and comparison groups)

* No significant medical history (ASA ≤ 2), syndromic conditions, cleft lip and/or palate.
* Have an existing (full) pan-oral radiograph at recruitment or subsequently undergoes one for routine diagnostic purposes.
* Child able to accept detailed clinical examination, radiographs (and photographs).
* Parents and child able to consent/assent to participate in the study and have sufficient level of literacy/understanding to complete written consent forms (with support if necessary).

MIH-group specific inclusion criteria.

* Children diagnosed with MIH by a specialist in paediatric dentistry according to validated diagnostic criteria (Ghanim et al., 2017, Ghanim et al., 2019) Comparison-group specific inclusion criteria
* Children referred to the host centre for the management of any dental condition other than MIH.

MIH-group specific exclusion criteria

* Children with an enamel defect that is not typical of MIH. Comparison-group specific exclusion criteria
* Children with an atypical pattern of dental caries/extraction in their first permanent molars such that a possible diagnosis of MIH could not be excluded (Ghanim et al., 2017, Ghanim et al., 2019).

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population is children referred to any of the participating paediatric dentistry clinics for assessment or treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1279 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
Prevalence of a dental anomaly in children with and without MIH | recruitment until July 2023
  Presence of any dental anomaly (number, shape, eruption disturbance)

SECONDARY OUTCOMES:
Characteristics associated with presence of a dental anomaly in children with MIH | recruitment until July 2023
  Secondary outcome measures for this study include the clinical and/or radiographic severity of MIH in relation to participants' gender, ethnicity/country and their global self-reported oral health,

CONTACTS AND LOCATIONS:
Overall Officials: Helen Rodd, BDS PhD, Principal Investigator — University of Sheffield
Locations (1):
- Charles Clifford Dental Hospital, Sheffield, S Yorks, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No participant data will be shared outside the core research team

REFERENCES:
- [Background] Walshaw EG, Noble F, Conville R, Anne Lawson J, Hasmun N, Rodd H. Molar incisor hypomineralisation and dental anomalies: A random or real association? Int J Paediatr Dent. 2020 May;30(3):342-348. doi: 10.1111/ipd.12601. Epub 2019 Dec 13. PMID 31790155
- [Background] Baccetti T. A controlled study of associated dental anomalies. Angle Orthod. 1998 Jun;68(3):267-74. doi: 10.1043/0003-3219(1998)0682.3.CO;2. PMID 9622764
- [Background] Brook AH. Variables and criteria in prevalence studies of dental anomalies of number, form and size. Community Dent Oral Epidemiol. 1975 Nov;3(6):288-93. doi: 10.1111/j.1600-0528.1975.tb00326.x. PMID 1104248
- [Background] Ghanim A, Silva MJ, Elfrink MEC, Lygidakis NA, Marino RJ, Weerheijm KL, Manton DJ. Molar incisor hypomineralisation (MIH) training manual for clinical field surveys and practice. Eur Arch Paediatr Dent. 2017 Aug;18(4):225-242. doi: 10.1007/s40368-017-0293-9. Epub 2017 Jul 18. PMID 28721667
- [Background] Schwendicke F, Elhennawy K, Reda S, Bekes K, Manton DJ, Krois J. Global burden of molar incisor hypomineralization. J Dent. 2018 Jan;68:10-18. doi: 10.1016/j.jdent.2017.12.002. Epub 2017 Dec 6. PMID 29221956